CLINICAL TRIAL: NCT07398118
Title: Treatment of Elderly Patients With Early Stage Breast Cancer (CRYO-1): The Efficacy of Cryoablation In The Elderly - A Phase II Multicentre, Feasibility Study.
Brief Title: CRYO-1: Cryoablation in Elderly Patients With Early-Stage Breast Cancer.
Acronym: CRYO-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Amphia Hospital (Other); Rijnstate Hospital (Other); Antoni van Leeuwenhoek Hospital (Other)
Responsible Party: Principal Investigator, Iza Stekelenburg, Coordinating investigator, St. Antonius Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R25.102
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Stage I; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Cryoablation; Early-stage breast cancer; Non-curative; Elderly; Minimally invasive treatment; Breast tumour; Local tumour control; Feasibility study; Cryotherapy; Non-surgical treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Intervention Model Description: This study uses a single-arm interventional model in which all participants undergo image-guided cryoablation as a one-time primary treatment. The study is designed to assess feasibility and safety in a selected population without randomisation or comparison to standard treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryoablation (Experimental): Participants receive image-guided percutaneous cryoablation as a single primary treatment for early-stage breast cancer. Cryoablation is performed to destroy the tumour by freezing, without surgical excision of the primary tumour.
  Interventions: Procedure: Cryoablation / Cryotherapy

INTERVENTIONS:
Procedure: Cryoablation / Cryotherapy — Cryoablation is performed as a percutaneous, image-guided procedure in which the breast tumour is destroyed by controlled freezing. One or more cryoprobes are placed into the tumour under imaging guidance, and freezing cycles are applied to achieve complete local tumour ablation. The procedure is performed as a single intervention without surgical excision of the primary tumour.

SUMMARY:
This study looks at a new way to treat early-stage breast cancer in older adults using a freezing technique called cryoablation.

Older adults with early-stage breast cancer are usually treated with surgery or primary endocrine therapy (hormone therapy). While these treatments can be effective, they may also be burdensome. Surgery can lead to pain, slow recovery, or complications, and primary endocrine therapy often requires long-term medication and may cause side effects or stop working over time. Cryoablation may offer a less invasive treatment option.

The goal of this study is to find out whether cryoablation can be safely and successfully used as the main treatment for older adults with early-stage breast cancer. Cryoablation destroys the tumour by freezing it. The procedure is performed through the skin using imaging guidance and does not involve surgical removal of the tumour.

Participants in this study are adults aged 70 years or older who have a small breast tumour that has not spread to the lymph nodes. All participants receive cryoablation as a single treatment.

After the procedure, participants are followed closely. Researchers will collect information on side effects, recovery, whether additional treatment is needed, and how participants experience the treatment. Quality of life will also be assessed.

This study is carried out in several hospitals. All participants must give written informed consent before taking part. The results of this study may help determine whether cryoablation could be a safe and practical treatment option for older adults with early-stage breast cancer and guide future research.

DETAILED DESCRIPTION:
CRYO-1 is a multicentre, phase II, single-arm interventional feasibility study evaluating cryoablation as a primary treatment for older adults with early-stage breast cancer. The study includes participants aged 70 years or older with clinically node-negative (cT1N0), estrogen receptor-positive, HER2-negative invasive breast cancer.

Standard treatment for this patient population consists of surgery or primary endocrine therapy. Although effective, both approaches may be associated with treatment burden in older adults. Surgical treatment may result in perioperative morbidity, while primary endocrine therapy requires prolonged treatment and may be associated with side effects and the development of endocrine resistance. Cryoablation is a minimally invasive, image-guided technique that induces tumour destruction by freezing and may reduce treatment burden in selected patients.

In this study, cryoablation is performed percutaneously under imaging guidance as a single procedure, without surgical excision of the primary tumour. The intervention is investigated as an alternative local treatment strategy in this selected population.

The primary objective of CRYO-1 is to assess feasibility and acute safety of cryoablation. Feasibility is defined by successful completion of the procedure, and safety is assessed by the incidence of treatment-related adverse events within three months, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

Secondary objectives include technical success, need for additional locoregional treatment, early local tumour control, patient tolerance, and health-related quality of life. Exploratory objectives include longer-term oncologic outcomes and identification of factors associated with successful local control.

CRYO-1 is an investigator-initiated study conducted across multiple hospitals. All participants provide written informed consent prior to enrolment. The study aims to generate prospective evidence on the feasibility and safety of cryoablation in older adults with early-stage breast cancer and to inform the design of future comparative or de-escalation studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Histologically confirmed invasive breast cancer
* Clinical stage cT1N0M0 based on mammography and ultrasound ER-positive, HER2-negative (IHC 0-1+ or 2+ with negative ISH), any PR status
* Presence of concurrent DCIS is allowed if limited to <25% of the pre-NST biopsy, with no radiologic suspicion of an extensive component
* Unifocal disease <2 cm, well visualized on ultrasound, with a minimum distance of ≥5 mm from the skin, nipple and thoracic wall
* Ability and willingness to comply with project requirements
* Preoperative endocrine therapy is allowed
* Written informed consent given by the subject

Exclusion Criteria:

* Pure DCIS lesions without invasive component
* Extensive calcifications on imaging suggestive of widespread disease
* Invasive lobular carcinoma (as assessed by IHC)
* Triple-negative or HER2-positive subtype (defined as (IHC 3+ or ISH positive)
* History of ipsilateral breast cancer or DCIS
* Prior ipsilateral radiotherapy
* Inability to communicate in Dutch or English language
* Planned (e)migration or long-term stay abroad within one year after inclusion

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Females
Enrollment: 61 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acute safety of cryoablation | Up to 6 months after cryoablation
  Feasibility is defined as successful completion of the cryoablation procedure as planned. Acute safety is assessed by the incidence of treatment-related adverse events following cryoablation, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
  Acute toxicity is graded according to the CTCAE v5.0 grading system, which classifies adverse events on an ordinal scale from Grade 1 (mild) to Grade 5 (death related to adverse event). The minimum score is Grade 1 and the maximum possible score is Grade 5. Higher grades indicate more severe toxicity (worse outcome).

SECONDARY OUTCOMES:
Technical success of cryoablation | During the cryoablation procedure
  Technical success is defined as correct placement of the cryoprobe(s) and completion of the planned freeze-thaw cycles resulting in complete coverage of the target tumour.
Local tumour control | Up to 12 months after cryoablation
  Local tumour control is defined as absence of residual or recurrent tumour at the treated site based on imaging and clinical follow-up.
Patient-reported tolerance and quality of life | Baseline and up to 12 months after cryoablation
  Participant-reported tolerance of the procedure and health-related quality of life assessed using validated questionnaires.
Need for additional locoregional treatment | Up to 12 months after cryoablation
  The proportion of participants requiring additional breast surgery or other locoregional treatment following cryoablation.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Amphia Hospital, Breda, North Brabant
  - Antoni van Leeuwenhoek - Nederlands Kanker Instituut, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive health information, and data sharing was not included in the informed consent or study protocol. Data will be analysed by the study team in accordance with applicable data protection regulations.